CLINICAL TRIAL: NCT00002838
Title: Phase I/II Pilot Study of Allogeneic Peripheral Blood Stem Cell Infusion For Patients With High Risk Chronic Lymphocytic Leukemia
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM95-194; P30CA016672 (NIH); MDA-DM-95194 (Other: UT MD Anderson Cancer Center); NCI-V96-1018; CDR0000065053 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia
Keywords: stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Chemotherapy + PSCT (Experimental): PSCT = Peripheral Stem Cell Transplantation
  Interventions: Biological: Filgrastim (G-CSF); Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: Filgrastim (G-CSF)
  Other Names: G-CSF; Neupogen
Drug: Cyclophosphamide
  Other Names: Cytoxan; Neosar
Drug: Fludarabine Phosphate
  Other Names: Fludara
Procedure: Peripheral Blood Stem Cell Transplantation
  Other Names: PBSCT; Stem Cell Transplant

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy and kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating patients with refractory chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility and toxicity of using allogeneic peripheral blood stem cell transplantation after intensive, but non-myeloablative chemotherapy with fludarabine/cyclophosphamide in patients with advanced chronic lymphocytic leukemia. II. Determine the engraftment kinetics and degree of chimerism available with this strategy.

OUTLINE: This is a nonrandomized, dose-seeking study. Stem cell donors receive G-CSF for 4 days prior to and throughout stem cell harvest. Patients receive intensive chemotherapy with fludarabine and cyclophosphamide for 3 days, with patients entered at increasing doses of both drugs until the dose allowing engraftment is determined. Three days after intensive chemotherapy, allogeneic stem cells are infused. Responding patients who do not experience worse than grade 1 acute graft-vs.-host disease receive additional stem cell infusions after 60 and 120 days. Patients are followed monthly for 4 months, at 6 and 12 months, then yearly for 5 years.

PROJECTED ACCRUAL: Up to 25 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Advanced chronic lymphocytic leukemia (Rai stage 3 or 4) with at least one of the following high-risk factors: Beta-2 microglobulin 3 or greater Abnormalities of chromosome 17 Other cytogenetic abnormalities Refractory to fludarabine-based chemotherapy or failure to achieve complete remission after 6 courses of a fludarabine-based regimen HLA-identical sibling donor willing and able to undergo apheresis for harvest of G-CSF-stimulated peripheral blood stem cells

PATIENT CHARACTERISTICS: Age: 65 and under Performance status: Zubrod 0 or 1 Hematopoietic: Not specified Hepatic: Bilirubin less than 1.5 mg/dL Renal: Creatinine less than 1.5 mg/dL Cardiovascular: No symptomatic cardiac disease Pulmonary: No symptomatic pulmonary disease Other: No active uncontrolled infection

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1995-12; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Feasibility + Toxicity of Combination Chemotherapy Plus Peripheral Stem Cell Transplantation | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Issa Khouri, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org